CLINICAL TRIAL: NCT02500563
Title: Exploratory/Proof of Principle Microbiota Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: Midwest Children's Health Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 6032
Record Dates: First submitted 2015-07-15; First posted 2015-07-16 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Fecal Microbiota

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amino acid based infant formula (Active Comparator)
  Interventions: Other: Amino acid based infant formula
- Extensively hydrolyzed casein infant formula (Experimental)
  Interventions: Other: Extensively hydrolyzed casein infant formula
- Mother's own breast milk (Other)
  Interventions: Other: Mother's own breast milk

INTERVENTIONS:
Other: Amino acid based infant formula
  Arms: Amino acid based infant formula
Other: Extensively hydrolyzed casein infant formula
  Arms: Extensively hydrolyzed casein infant formula
Other: Mother's own breast milk
  Arms: Mother's own breast milk

SUMMARY:
This clinical trial will evaluate the stool of infants fed one of two infant formulas, which contain different types of proteins, or breast milk to determine if different proteins have an effect on the type of bacteria that enters and lives in an infant's intestine early in life.

DETAILED DESCRIPTION:
This clinical trial will evaluate the stool of infants fed one of two infant formulas, which contain different types of proteins, or breast milk to determine if different proteins have an effect on the type of bacteria that enters and lives in an infant's intestine early in life.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, 1-7 days of age at registration or randomization
* Term infant with appropriate birth weight for gestational age
* Either solely formula fed or exclusively receiving mother's own breast milk
* Signed Informed Consent and Protected Health Information

Exclusion Criteria:

* Caesarean delivery
* Infant was born from a mother with Type 1 diabetes
* History of underlying metabolic or chronic disease or immunocompromised
* Feeding difficulties or history of formula or human milk intolerance
* Signs of acute infection of current use of antibiotics

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota measured at each visit | 8 weeks
  Sequencing and composition of samples

SECONDARY OUTCOMES:
Body weight measured at each visit | 8 weeks
  Measurement collected with a calibrated infant scale
Body length measured at each visit | 8 weeks
  Measurement collected with a standardized length board
Head circumference measured at each visit | 8 weeks
  Measurement collected with a standardized measuring tape
Parental recall of formula intake at each visit | 8 weeks
Stool collection at each visit | 8 weeks
  Composite measure of pH and short chain fatty acids
Serious adverse events collected throughout the study period | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jon Vanderhoof, M.D., Study Director — Mead Johnson and Company
Locations (1):
- Midwest Children's Health Research Institue, Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Kok CR, Brabec B, Chichlowski M, Harris CL, Moore N, Wampler JL, Vanderhoof J, Rose D, Hutkins R. Stool microbiome, pH and short/branched chain fatty acids in infants receiving extensively hydrolyzed formula, amino acid formula, or human milk through two months of age. BMC Microbiol. 2020 Nov 9;20(1):337. doi: 10.1186/s12866-020-01991-5. PMID 33167908
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765